CLINICAL TRIAL: NCT03294551
Title: Enhancing HPV Vaccination Rates for 11-14 Year Old Adolescents Using New York State's Immunization Information System
Brief Title: HPV Centralized R/R RCT #2 - New York State
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Colorado, Denver (Other); New York State Department of Health (Other Government)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Vice Chair Clinical Research, Pediatrics, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17-001559; 5R01CA187707-02 (NIH)
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Vaccines
Keywords: HPV Vaccine; immunization registry; Reminder recall (R/R)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care Control (No Intervention): Usual source of care
- HPV Vaccine Reminder Recall - Autodialer (Experimental): HPV Vaccine Reminder Recall - Autodialer: Receive up to 4 reminders via telephone (live call or voicemail) - includes brief educational message + providers name + providers telephone number
  Interventions: Behavioral: HPV Vaccine Reminder Recall - Autodialer
- HPV Vaccine Reminder Recall - Texting (Experimental): HPV Vaccine Reminder Recall - Texting: Receive up to 4 reminders via text message - includes brief educational message + providers name + providers telephone number
  Interventions: Behavioral: HPV Vaccine Reminder Recall - Texting

INTERVENTIONS:
Behavioral: HPV Vaccine Reminder Recall - Autodialer — Investigators will send out HPV vaccine reminder recall notices via autodialer message to the parents of adolescents 11-14 years of age who are eligible to receive a dose of the HPV vaccine per the records in the New York State Immunization Information System (NYSIIS). The investigators will be testing the effectiveness and cost effectiveness of the various modalities or reminders as compared to the standard of care control (no reminders)
  Arms: HPV Vaccine Reminder Recall - Autodialer
Behavioral: HPV Vaccine Reminder Recall - Texting — Investigators will send out HPV vaccine reminder recall notices via text message to the parents of adolescents 11-14 years of age who are eligible to receive a dose of the HPV vaccine per the records in the New York State Immunization Information System (NYSIIS). The investigators will be testing the effectiveness and cost effectiveness of the various modalities or reminders as compared to the standard of care control (no reminders)
  Arms: HPV Vaccine Reminder Recall - Texting

SUMMARY:
The work done in this trial builds off of the work previously conducted by this same research group in clinicaltrials.gov ID: NCT03057379. Due to some changes in study design, protocol, and cohort of interest, a new registration was warranted.

The overarching goal of this study is to evaluate the effectiveness, cost-effectiveness, and sustainability of utilizing statewide immunization information systems (IISs) to conduct centralized reminder recall (R/R) to improve human papillomavirus (HPV) vaccination rates among adolescents 11-14 years of age.

The latest recommendations from the ACIP, as of February 2017, modified the vaccination schedule for the HPV series for eligible adolescents ages 11-14. Adolescents who receive dose #1 between the ages of 11 and 14 are now eligible for their second and final dose 6-12 months after their initial dose. Despite U.S. guidelines for vaccinating all adolescents starting at age 11 with the HPV vaccine, in 2012 only 53% of 13-17 year old females had >1 dose and 35% had 3 doses; 21% of teen males had a vaccination. Modeling studies predict marked reduction in HPV associated cancers and in disparities in these cancers if high HPV vaccination rates can be achieved.

With this new dosing schedule for adolescents, the research team proposes to conduct a randomized control trial (RCT) utilizing the capabilities of the State Immunization Information System (IIS), and create a HPV-specific R/R autodialer and text message to be delivered to the parents of patients ages 11-14 of randomly selected practices within New York State (excluding NYC). Upon conclusion of this trial, researchers will develop a toolkit for dissemination so that other state IIS systems may replicate these centralized reminder recall procedures.

DETAILED DESCRIPTION:
The overarching goal is to evaluate the effectiveness, cost effectiveness, and sustainability of statewide immunization systems (IISs) to conduct reminder/recall (R/R) to improve human papillomarvirus (HPV) vaccination rates among adolescents ages 11-14.

Each year, 6.2 million persons are newly infected with HPV and 26,000 new HPV-related cervical, genital, and oropharyngeal cancers are diagnosed, resulting in >$4 billion in annual medical costs. Despite U.S. guidelines for vaccinating all adolescents starting at age 11 with the HPV vaccine, in 2012 only 53% of 13-17 year old females had >1 dose and 35% had 3 doses; 21% of teen males had a vaccination.

The most effective strategy for improving vaccination rates is patient reminder/recall (R/R). Recent literature from Melissa Stockwell found that utilization of a new R/R modality, i.e. text messaging, positively impacted influenza vaccination rates among the adolescents enrolled in the study. Although R/R is already considered a "best practice" for improving vaccination rates, very few practices use reminder/recall for any vaccinations because of costs and lack of personnel time; and even fewer use reminder/recall for HPV vaccine.

Furthermore, since the Advisory Committee on Immunization Practices (ACIP) modified the schedule for the HPV series for adolescents' age 11-14 years, those who receive dose #1 between ages of 11 and 14 years are now eligible for their second and final dose 6-12 months after their initial dose. This change in dosing schedule could influence HPV vaccine visit scheduling procedures within Family Practice and/or Pediatric Clinics, and would therefore effect timing and frequency of any R/R strategies currently in place. Therefore, the UCLA (overseeing the work to be done in NY) and University of Colorado at Denver research teams unite to understand how the use of centralized R/R to disseminate reminders, via text messages and autodialer calls, to patients eligible for the 2-dose HPV vaccine could impact vaccination rates among adolescents ages 11-14. This will be the first head-to-head RCT comparing text message vs. autodialer reminders to standard of care control

The aim of the study is as follows:

To assess the impact and cost-effectiveness of autodialer IIS R/R versus text message based IIS R/R versus standard-of-care control (no reminder recall) in increasing initiation and completion of the 2-dose HPV vaccine series among adolescents 11-14 years of age. The investigators will use a within-practice randomized control trial, randomizing patients within 150 practices to the aforementioned intervention arms.

Hypothesis 1: All centralized IIS R/R modalities will be more effective than usual care

Hypothesis 2: Text messaging will be more cost-effective than other modalities

Upon completion of the study, the investigators will have a feasible, sustainable, cost-effective model for HPV vaccination reminders that could be scaled up on the national level to help prevent HPV-related cancers. Additionally, this research will be adding significant new knowledge to the field as no such studies exist examining the impact of educational text message R/R on HPV vaccination rates among adolescents eligible for the 2-dose series.

ELIGIBILITY:
Inclusion Criteria:

* 11 to 14 years of age
* patient of a participating practice in New York State (practices were randomly selected)
* is due for an HPV dose at baseline, or
* has initiated but not yet completed the HPV series at baseline
* immunization record within the New York State Immunization Information System (NYSIIS) database

Exclusion Criteria:

* is not a patient of a participating practice that was randomly selected in New York State
* has completed the HPV vaccination series
* does not have a valid record within the NYSIIS database

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37003 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Initiation of the HPV 2-dose series | 5 months from the first reminder received for the first dose of HPV vaccine
  Receipt and documentation of the initial dose of the vaccine within the series as recorded in the NYSIIS database. Investigators are allowing 5 months after the initial reminder recall was sent as the timeline of attributing vaccination status to the intervention
Completion of the HPV 2-dose series | 5 months from the first reminder received for the last dose of HPV vaccine
  Receipt and documentation of the final dose of the vaccine series as recorded within the NYSIIS database. Investigators are allowing up to 5 months after the first reminder recall for the second dose was received. If vaccination is received after that 5 month period, investigators will not attribute change in vaccination status to the reminder.

SECONDARY OUTCOMES:
Cost of the R/R intervention - autodialers and texting | 17 months - entirety of the trial
  A cost-effectiveness analysis will be conducted to determine which modality of R/R (autodialer or text message) is the most cost-effective in relation to improving HPV vaccination rates among 11-14 year old adolescents as compared to the control, as well as comparing the two interventions arms to one another.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szilagyi, MD MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
The aggregate results will be published in a peer reviewed journal.

REFERENCES:
- [Derived] Gurfinkel D, Kempe A, Albertin C, Breck A, Zhou X, Vangala S, Beaty B, Rice J, Tseng CH, Campbell JD, Valderrama R, Rand C, Humiston SG, Roth H, Arora S, Szilagyi P. Centralized Reminder/Recall for Human Papillomavirus Vaccination: Findings From Two States-A Randomized Clinical Trial. J Adolesc Health. 2021 Oct;69(4):579-587. doi: 10.1016/j.jadohealth.2021.02.023. Epub 2021 Apr 10. PMID 33846054